CLINICAL TRIAL: NCT04711278
Title: Hypnosis Mask in Pre-operative Anxiety Management in Ambulatory Surgery Patients: Using Virtual Reality
Brief Title: Using Virtual Reality to Prevent Pre-operative Anxiety in Ambulatory Surgery Patients
Acronym: PACAH-UCA HV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP201445; 2019-A03316-51 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-01-07; First posted 2021-01-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-11

CONDITIONS: Hallux Valgus; Surgery
Keywords: hallux valgus; hypnosis; pre-operative anxiety; surgery
MeSH Terms: conditions — Hallux Valgus | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypnosis group (Experimental): Mask-wearing as hypnosis method for patients in this arm.
  Interventions: Device: Mask-wearing hypnosis
- comparator group (Sham Comparator): No hypnosis for patients in this arm.
  Interventions: Other: Without hypnosis

INTERVENTIONS:
Device: Mask-wearing hypnosis — Virtual mask will be worn by patients before and during surgery of Hallux valgus to realize hypnosis.
  Virtual mask with 2 types of voice: female voice and male voice. Several types of image or music to choice by patient.
  Arms: hypnosis group
Other: Without hypnosis — No hypnosis during surgery of Hallux valgus.
  Arms: comparator group

SUMMARY:
The primary objective is to evaluate the impact on pre-operative anxiety management of using the virtual reality mask for surgery of hallux valgus.

DETAILED DESCRIPTION:
As secondary objectives, the study aims

* to evaluate post-operative analgesic according to non-drug pre-operative hypnosis, measured by reduction in analgesic intake, and by evaluate of pain;
* to evaluate factors which permitting discharge rapidly from hospital in case of hypnosis with virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years;
* Autonomous patient living at home;
* Affiliated to a social security scheme;
* Informed consent signed by patient;
* Patient will undergo a planned ambulatory surgery for hallux valgus.

Exclusion Criteria:

* Inability to understand STAI-A questionnaire;
* Patient refusal;
* Patient underwent a bilateral surgery;
* Patient judicial decision;
* Covered by french AME health system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Anxiety assessment at baseline | baseline, pre-intervention
  The State Trait Anxiety Inventory (STAI) will be used to measure anxiety levels.
Anxiety assessment after the surgery | immediately after the surgery
  The State Trait Anxiety Inventory (STAI) will be used to measure anxiety levels.

SECONDARY OUTCOMES:
Analgesic taken | at the end of study, an average of 1 day
  Dose of analgesic taken will be added up.
Duration of stay | at the end of study, an average of 1 day
  Duration of stay before discharge of hospital.
Pain assessment | day 1
  EVA score, a french auto evaluation tool will be used for pain.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MENIGAUX, MD, Principal Investigator — Department of Orthopaedics and Traumatology, Ambroise Paré hospital, APHP; Marie-Hélène SANDIFORD, Study Director — Department of Orthopaedics and Traumatology, Ambroise Paré hospital, APHP
Locations (1):
- Department of Orthopaedics and Traumatology, Ambroise Paré hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganry L, Hersant B, Sidahmed-Mezi M, Dhonneur G, Meningaud JP. Using virtual reality to control preoperative anxiety in ambulatory surgery patients: A pilot study in maxillofacial and plastic surgery. J Stomatol Oral Maxillofac Surg. 2018 Sep;119(4):257-261. doi: 10.1016/j.jormas.2017.12.010. Epub 2018 Jan 6. PMID 29317347